CLINICAL TRIAL: NCT03512639
Title: Arnica Montana and Bellis Perennis for Prevention of Seroma Following Mastectomy and Immediate Breast Reconstruction: Prospective, Randomized, Double-Blind, Placebo- Controlled Trial
Brief Title: Arnica Montana and Bellis Perennis for Prevention of Seroma After Mastectomy
Acronym: HOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0136-16
Record Dates: First submitted 2018-04-09; First posted 2018-05-01 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2016-06

CONDITIONS: Seroma
Keywords: Mastectomy, Breast Reconstruction, Homeopathic Treatment
MeSH Terms: conditions — Seroma | interventions — Arnicae flos extract

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider, Investigator
Masking Description: The medications were packed in bottles, each containing 5 grams of the preparation, and consecutively numbered. The prefix 'A' indicated Arnica montana, and 'B' Bellis perennis .
  Participants were randomly allocated into groups given either homeopathic medication (Arnica montana C30 and Bellis perennis C30) or placebo (alcohol 40% and alcohol 40%) in a 1:1 ratio. . The randomization code was held in confidence and the code was not broken until the data analysis. The same randomization list was used to blind the Arnica montana and the Bellis perennis, creating similar pairs. The placebos and the active medication were indistinguishable in appearance, taste and smell.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Active Comparator): Patients in the study group were given homeopathic medication (Arnica montana C30 and Bellis perennis C30) .
  Interventions: Drug: Homeopathic Medication
- control (Placebo Comparator): Patients in the control group were given placebo medication. The placebos and the active medication were indistinguishable in appearance, taste and smell
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Homeopathic Medication — Homeopathic medication (Arnica montana and the Bellis perennis) were given to women in the study group following mastectomy and reconstruction to reduce post operative seroma
  Other Names: Arnica montana and the Bellis perennis
  Arms: Study
Drug: Placebo — placebo was given to women in the control group following mastectomy and reconstruction to reduce post operative seroma
  Arms: control

SUMMARY:
Arnica montana and Bellis perennis for Prevention of Seroma Following Mastectomy.

DETAILED DESCRIPTION:
Background Seroma is a common surgical complication created by the inflammatory process that follows mastectomy and reconstruction. It is, thus, common practice to insert surgical drains, which often often remain in place for long periods and delay recovery. In light of the many advantages of holistic treatment, there has been a global trend of integrating them with conventional medicine. In this study, the investigators examined the effect of Arnica montana and Bellis perennis on seroma prevention after mastectomy and breast reconstruction.

Study design The investigators conducted a prospective, double-blind, randomized, controlled study to asses the effect of homeopathic remedies on seroma in 55 patients (78 breasts), who had undergone mastectomy for cancer or risk reduction, followed by immediate implant and Acellular Dermal Matrix (ADM)-based breast reconstruction in the Department of Plastic & Reconstructive Surgery at Shaare Zedek Medical Center in Jerusalem, Israel, between January 2016 and August 2017 (Figure 1). The study protocol was approved by the Institutional Review Board and it was registered on the ClinicalTrials.gov register.

Subjects All subjects were female, aged over 18 years, who underwent mastectomy, either for breast cancer or for risk reduction, followed by immediate breast reconstruction. In some patients, this was performed in a single procedure - direct to implant (DTI) (n=42); in others, it was in two stages tissue expander (TE) (n=36), depending on presurgical evaluation, risk factors and clinical assessment of perfusion of the mastectomy skin flaps. All subjects signed informed consent forms after receiving a detailed explanation of the study from one of its investigators.

The investigators excluded patients with: (a) conditions which could affect wound-healing; (b) coagulation problems (autoimmune and hematological diseases, etc.); (c) taking medication which affects the immunological or hematological system (steroids, anticoagulants, chemotherapeutic agents, etc.); and (d) with unbalanced background diseases. Active smokers were instructed to stop smoking at least three weeks prior to surgery and a month postoperatively.

Study medication and randomization and surgical techniques Experimental medications and placebos were prepared and delivered in accordance with the Homeopathic Pharmacopoeia of the United States (HPUS). Stem tinctures of Arnica montana, Bellis perennis and 40% alcohol as placebo were diluted 1:100 with 40% alcohol, and vigorously shaken. This process was repeated 30 times for a theoretical final concentration of 10-60 of the stem solutions. Spherical saccharose globules, approximately 1 mm in diameter, were wetted with the diluted tinctures and dried, resulting in three groups of the experimental medication: Arnica montana C30 (10-60), Bellis perennis C30 (10-60) and alcohol dilutions as placebo. The medications were packed in bottles, each containing 5 grams of the preparation, and consecutively numbered. The prefix 'A' indicated Arnica montana, and 'B' Bellis perennis .

Participants were randomly allocated into groups given either homeopathic medication (Arnica montana C30 and Bellis perennis C30) or placebo (alcohol 40% and alcohol 40%) in a 1:1 ratio. Age, body mass index, laterality of mastectomy, mastectomy type and number requiring sentinel lymph node biopsy and axillary dissection were similar between groups. The randomization sequence was created by an independent physician, uninvolved in the study, using computer-generated random numbers. The randomization code was held in confidence and the code was not broken until the data analysis. The same randomization list was used to blind the Arnica montana and the Bellis perennis, creating similar pairs. The placebos and the active medication were indistinguishable in appearance, taste and smell. Three globules of each medication were regarded as a single dose, to be sucked rather than swallowed.

Patients were hospitalized the night prior to surgery. On admission, a member of the study team again explained the study protocol, and gave the assigned medications to the patients. Patients were asked to take the medication according to the following protocol (Figure 2):

1. One dose of A (3 pills) on the morning of surgery.
2. One dose of A and one of B, 4 to 6 times a day for the first 24 hours after surgery (as soon as patients were stable, conscious and nausea- and vomit-free).
3. One dose of A and one of B, 3 times a day until 4 days after surgery.
4. Finally, one dose of B 3 times a day until removal of the surgical drain. All mastectomies were performed by experienced breast surgeons at our institution. Amputated breast-weight was documented. Sentinel lymph-node biopsy (SLNB) or axillary lymph-node dissection (ALND) was carried out according to the oncological status of each patient, either through a separate axillary incision or through the mastectomy incision. All reconstructions were subpectoral ADM-assisted, performed by plastic surgeons from our department. 42 breasts underwent the DTI procedure, and in 36 breasts a two-stage TE approach was taken, according to the patient's estimated breast volume, risk factors and intraoperative clinical evaluation of flap perfusion. ADM used was an 8*16 cm ADM. A 10-mm Jackson-Pratt drain was inserted through a subcutaneous tunnel in the lateral breast gutter at the level of the inframammary fold (IMF) (in the subcutaneous space). When axillary lymph node dissection (ALND) was performed through a separate incision, a second drain was placed in the axillary space. Drains were removed when drainage fell below 30 mL/24 hours.

Assessment

The following data for all patients were retrieved from their medical records:

* Baseline characteristics and demographic variables
* Medical history and risk factors - comorbidities, obesity, smoking, breast cancer (BRCA) mutation status
* Variables relating to the procedure - reason for surgery (breast cancer vs. risk reduction), breasts operated (unilateral or bilateral), size and type of implant (DTI vs. TE and implant volume) and lymph node status (no biopsy taken/sentinel lymph node biopsy (SLNB)/ALND)
* Postoperative course- time to drain removal, hemoglobin and cortisol levels on postoperative days (POD) 3 and 7, postoperative level of pain according to the visual analog (VAS) scale and Quality of Recovery. The VAS scale is a scale from 0 to 10, with 0 being "no pain at all" and 10 being "worst pain imaginable." The staff nurse caring for each patient administered the form and elicited the patient response for pain level according to the study protocol, and the quantity of narcotics taken. On POD 3 and 7, patients were given the Quality Of Recovery (QoR) 40 questionnaire, a validated questionnaire to measure postsurgical quality of recovery. Its scores range from 40 for very poor recovery to 200 for outstanding quality of recovery [49-51].
* Postoperative complications: hematoma, skin-flap necrosis, infection, seroma, explantation and need for repeat surgery. Complications were divided into major and minor. Major complications included any of those mentioned above which required revision surgery in the operating room. Minor complications resolved spontaneously or were treated at the bedside.

Data analysis All data were collected daily by a study coordinator. The investigators calculated the mean standard deviation (SD) and range for all quantitative variables, as well as their absolute frequencies and percentages. Statistical analyses were conducted using statistical software. The criterion for significance was: alpha (α) = .05 (one-sided).

ELIGIBILITY:
Inclusion Criteria:

* Female patients, aged over 18 years.
* Patients underwent mastectomy, either for breast cancer or for risk reduction, followed by immediate breast reconstruction.
* All subjects signed informed consent forms. -

Exclusion Criteria:

* Conditions which could affect wound-healing
* Coagulation problems (autoimmune and hematological diseases, etc.)
* Medication which affects the immunological or hematological system (steroids, anticoagulants, chemotherapeutic agents, etc.)
* Unbalanced background diseases.
* Active smokers were instructed to stop smoking at least three weeks prior to surgery and a month postoperatively.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 55 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Reduction of post operative seroma following mastectomy and reconstruction. | 18 months
  Evaluate the effect of Arnica montana and Bellis perennis on seroma formation, measured in number of days to surgical drain removal, in patients undergoing mastectomy and reconstruction.

IPD SHARING:
Plan to Share IPD: No